CLINICAL TRIAL: NCT02891330
Title: Assessing the Impact of an Educational Personalized Clinical Support Device Preventive and a Referent Nurse in Surgery for Obesity With the Risk of Occurrence of Dumping Syndrome After Gastric Bypass.
Brief Title: Impact of an Educational Personalized Clinical Support Device Preventive and a Referent Nurse in Surgery for Obesity
Acronym: IRCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014_17; 2015-A00646-43 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Dumping Syndrome
Keywords: Roux-en-Y Gastric ByPass
MeSH Terms: conditions — Dumping Syndrome | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary and nutritional recommendations (Experimental): Postoperative personalized approach based on dietary and nutritional recommendations conducted by a nurse
  Interventions: Behavioral: Dietary and nutritional recommendations conducted by a nurse
- Standard of care (No Intervention): Postoperative standard of care

INTERVENTIONS:
Behavioral: Dietary and nutritional recommendations conducted by a nurse — Supplementary dietary and nutritional education
  Arms: Dietary and nutritional recommendations

SUMMARY:
The postprandial dumping syndrome is a frequent consequence of Roux-en-Y Gastric ByPass due to the rapid emptying of the stomach remnant in to the intestinal lumen. Dumping-related symptoms occur very early after eating (within 30 minutes), are not associated with concurrent hypoglycemia, and are most prominent in the early postoperative period. This syndrome very debilitating for the patient can be improved by dietary and nutritional recommendations. We hypothesize that a personalized approach based on dietary and nutritional recommendations conducted by a nurse would likely to decrease the frequency of dumping syndrome and improve the postoperative quality of life of patients in the early postoperative period.

DETAILED DESCRIPTION:
The Roux-en-Y Gastric ByPass is considered the gold standard of weight loss surgery and is the most commonly performed bariatric procedure worldwide.The postprandial dumping syndrome is a frequent consequence of gastrojejunal anastomosis due to the rapid emptying of the stomach remnant in to the intestinal lumen. Dumping-related symptoms occur very early after eating (within 30 minutes), are not associated with concurrent hypoglycemia, and are most prominent in the early postoperative period. The symptoms of dumping syndrome include nausea, abdominal cramps, diarrhea, dizzy spells, weakness and cold sweats either with or after eating.This syndrome very debilitating for the patient can be improved by dietary and nutritional recommendations. We hypothesize that an individualized approach based on dietary and nutritional recommendations and monitoring of patients conducted by a nurse in the first three months after surgery would likely to decrease these problems and improve the postoperative quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index ≥40 kg / m2 or ≥35 kg / m2 in the presence of comorbidities related to obesity
* Indication to Roux-en-Y Gastric ByPass

Exclusion Criteria:

* Contraindication to Roux-en-Y Gastric ByPass
* Refusal to sign the consent form
* Patient not affiliated to a social security system
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
The frequency of dumping syndrome | 3 months
  The frequency of dumping syndrome at 3 months will be compared between the two groups.

SECONDARY OUTCOMES:
Change in Body Mass Index | 3 months
Frequence of Adverse Events after surgery | at 1 and 3 months
Quality of Life-Lite questionnaire | 3 months
  Estimation of quality of life by Impact of Weight on Quality of Life-Lite questionnaire(IWQOL-Lite)
Personal Effectiveness Assessment questionnaire (SEPOB) | 3 months
  Measure the efficacy of therapeutic education by personal estimation of the level of skill using a specific obesity assessment questionnaire (SEPOB questionnaire or survey emotional, cognitive and behavioral sense of personal efficacy)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène VERKINDT, MD, Principal Investigator — University Hospital, Lille
Locations (4):
- France (4):
  - CH ARRAS, Arras
  - Ch Boulogne-Sur-Mer, Boulogne-sur-Mer
  - Hôpital Claude Huriez, CHRU, Lille
  - Ch de Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No